CLINICAL TRIAL: NCT05431062
Title: Comparison of US-guided Single-dose Thoracic Paravertebral Block, Erector Spinae Plane Block and Serratus Anterior Plane Block in Pediatric Patients Undergoing Thoracic Surgery.
Brief Title: Comparison of US-guided Single-dose Thoracic Paravertebral, Erector Spinae Plane and Serratus Anterior Plane Blocks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, associated professor, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2021/808
Record Dates: First submitted 2022-06-10; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia, Local
Keywords: thoracic paravertebral block; erector spinae plane block; serratus anterior plane block; ultrasound-guided; thorocotomy pain
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Prospective Observational Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic paravertebral block (Active Comparator): USG guided TPVB will be performed with 0.5 mL/kg %0.25 Buvicaine in the paravertebral space.
  Interventions: Drug: Bupivacain
- Erector spinae plane block (Active Comparator): USG guided ESPB will be performed with 0.5 mL/kg %0.25 Buvicaine into the facial plane between erector spine muscle and transverse process
  Interventions: Drug: Bupivacain
- Serratus anterior plane block (Active Comparator): USG guided ESPB will be performed with 0.5 mL/kg %0.25 Buvicaine into the facial plane between serratus anterior muscle and external intercostal muscles
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — %0.25
  Other Names: Marcaine

SUMMARY:
This study evaluates the analgesic effects of ultrasound-guided regional techniques, Thoracic Paravertebral Block (TPVB), Erector Spinae Plane Block (ESPB) and Serratus Anterior Plane Block(SAPB) by comparing postoperative total morphine consumption, first analgesic requirement time, and postoperative pain scores ( FLACC/NRS), postoperative chronic pain in 3rd month in pediatric patients undergoing thoracic surgery. The investigators also aim to observe the side effects of these techniques such as nausea, vomiting, bradycardia, hypotension, respiratory depression

DETAILED DESCRIPTION:
Thoracic surgery is one of the most common causes of postoperative severe pain due to the damage to intercostal nerves, irritation of the pleura and rib retraction. Effective analgesia provides patient comfort and enables early mobilization, reducing complications such as pneumonia, respiratory failure, hypoxia, and hypercapnia. In pediatric patients, nonsteroid anti-inflammatory drugs, opioids and regional analgesia techniques can be used for multimodal analgesia. Several side effects of opiates such as respiratory depression, nausea, vomiting, itching, addiction, and sedation effect patients' comfort and delay discharge. Nowadays US-guided truncal block techniques such as thoracic paravertebral block (TPVB) become popular. TPVB provide the somatosensorial and visceral block with an injection of the local anaesthetic agent into the paravertebral space. Existing evidence demonstrates the non inferiority of TPVB compared with TEA for postoperative analgesia and TPVB can reduce side effects. Erector Spina Plan Block (ESPB) was first described in 2016 as an ultrasound-guided truncal block for thoracic neuropathic pain and now ESPB uses for many different thoracics and abdominal surgeries for postoperative analgesia. Several studies have shown that ESPB can provide adequate analgesia in postoperative thoracic pain. ESPB is gaining popularity because its application is easy and safe compared with TPVB. Another new US-guided regional anaesthetic block technique, the serratus anterior plane block (SAPB), targets the plane above or below the serratus anterior muscle in the midaxillary line and provides analgesia to a hemithorax by blocking the lateral branches of the intercostal nerves, thoracicus longus and thoracodorsal nerves. The SAP block provides analgesia to the 2nd and 9th thoracic dermatomes. The SAP block is safe, and easy to perform, owing to its easy-to-learn technique and distinct bony landmarks. So, it can be an attractive alternative for pain relief after thoracic surgery.

In this study, Investigators aim to compare the efficacy of these three techniques in pediatric patients. The primary hypothesis is the analgesic efficacy of SAPB will be equivalent to TPVB and RSPB. The primer outcome is postoperative total narcotic analgesic consumption in 24 hours. The seconder outcomes are; time of postoperative first analgesic requirement, postoperative pain scores (FLACC - NRS) in 0.-15.-30.-45.minutes and 1.-2.-6.-12.-24.-48. hours, chronic thoracic pain 3 months after surgery, intraoperative additional fentanyl requirement, postoperative additional paracetamol requirement, intraoperative hemodynamic parameters, first mobilization time, side effects, technical complications, and the satisfaction of patient-surgeon.

ELIGIBILITY:
Inclusion Criteria:

1-14 age patients undergoing thoracic surgery, ASA 1-2-3, Patients without chronic opioid use

Exclusion Criteria:

Denial of patient or parents, Infection of the local anaesthetic area, Infection of the central nervous system, Coagulopathy, Brain tumours, Known allergy against local anaesthetics.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Iv Morphine Consumption | Up to 24 hours
  The total dosage of iv morphine consumption in 24 hours.

SECONDARY OUTCOMES:
Face, Legs Avtivity, Cry, Consolability (FLACC) scores | Up to 48 hours
  It corporates five categories of behavior, each scored on 0-2 point scale so that total score ranges from 0 to 10. Total scores of 0-3 is defined as mild or no pain, 4-7 as moderate, and 8-10 as severe pain
Postoperative NRS Score (Numeric Rating Scale) | Up to 48 hours
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Time of Postoperative First Analgesic Requirement Time | Up to 48 hours
  Time of postoperative first analgesic requirement time.
Additional IV Paracetamol Dosage In The Postoperative Period | Up to 48 hours
  15mg/kg iv paracetamol will be administered 30 minutes before extubation. In the postoperative follow-up that will be performed every 6 hours,15mg/kg iv paracetamol will be administered if the FLACC score is >3 or the NRS score is >4.
Intraoperative Heart Rate (beat/min) | Intraoperative Period
  To be measured through the operation at intervals of 5 minutes
Intraoperative Mean Arterial Pressure(MAP)(mmHg) | Up to end of the operation
  To be measured through the operation at intervals of 5 minutes
Number of patients who need intraoperative additional Fentanyl | Up to end of the operation
  Intraoperative Additional Fentanyl Requirement
Chronic Thoracic Pain | Up to 3 months
  Presence of thoracic pain due to the incision after 3 months of the thoracic surgery.
Length of Hospital Stay | Up to first week
  Length of Hospital Stay

OTHER OUTCOMES:
Incidence of PONV (postoperative nausea and vomiting) | Up to 48 hours
  Incidence of postoperative nausea and vomiting.
Respiratuar Depression | Up to 48 hours
  Incidence of respiratory depression due to ıv morphine in the postoperative follow-up.
Postoperative sedation scale | Up to 48 hours
  A numerical rating sedation scale requires the patient to rate their sedation on a defined scale. For example, 1: deeply asleep, 2: lightly asleep, 3: drowsy, 4: fully awake and alert
Itching | Up to 48 hours
  Incidence of itching due to iv morphine in the postoperative follow-up.
Incidence of Complications Due To The Regional Block | Up to first week
  Incidence of dural puncture,pneumothorax,infection,neural damage.
First Mobilization Time | Up to 48 hours
  First mobilization time .
Need of Intensive Care Unit Follow-Up | Up to 48 hours
  The number of patients who need ICU follow-up.
Family Satisfaction | Up to 48 hours
  Satisfaction score; 0: very unsatisfied 3:very unsatisfied
Surgeon Satisfaction | Up to 48 hours
  Satisfaction score; 0: very unsatisfied 3:very unsatisfied

IPD SHARING:
Plan to Share IPD: Undecided